CLINICAL TRIAL: NCT03081598
Title: A Phase 2, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of PBI-4050 in Type 2 Diabetes Mellitus Patients With Metabolic Syndrome
Brief Title: Study to Evaluate Safety, Efficacy of PBI-4050 & Its Effect on Relevant Biomarkers in T2DM Patients With Metabolic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to meet recruitment target during the recruitment period
Sponsor: Liminal BioSciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBI-4050-CT-9-08
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Type 2 Diabetes Mellitus; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — setogepram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Daily dose of 6 capsules of placebo
  Interventions: Other: Placebo
- PBI-4050 400 mg (Active Comparator): Daily dose of 2 capsules of PBI-4050 and 4 capsules of placebo
  Interventions: Drug: PBI-4050; Other: Placebo
- PBI-4050 800 mg (Active Comparator): Daily dose of 4 capsules of PBI-4050 and 2 capsules of placebo
  Interventions: Drug: PBI-4050; Other: Placebo
- PBI-4050 1200 mg (Active Comparator): Daily dose of 6 capsules of PBI-4050
  Interventions: Drug: PBI-4050

INTERVENTIONS:
Drug: PBI-4050 — Soft gelatine capsule containing 200 mg of the active ingredient per capsule
  Arms: PBI-4050 1200 mg; PBI-4050 400 mg; PBI-4050 800 mg
Other: Placebo — Placebo soft gelatine capsule
  Arms: PBI-4050 400 mg; PBI-4050 800 mg; Placebo

SUMMARY:
This is a Phase 2, multi-center, double-blind, placebo-controlled study of the safety and effect of PBI-4050 at doses ranging from 400 mg to 1200 mg on relevant biomarkers in subjects with inadequately-controlled T2DMS on stable background antidiabetic therapy.

DETAILED DESCRIPTION:
This Phase 2 study will be performed by 15 sites in Canada. The total duration of study participation for each subject is approximately 20 weeks and comprises 6 study visits

A total of approximately 268 subjects will be enrolled in the study and randomly assigned to one of the following 4 treatment groups:

* PBI-4050 400 mg
* PBI-4050 800 mg
* PBI-4050 1200 mg
* Placebo

All subjects will receive the assigned study drug for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older.
2. Subject has signed written informed consent.
3. Subject has a clinical diagnosis of T2DM with an HbA1c level between ≥ 7.5% and ≤ 10%.
4. Subject has been receiving stable antidiabetic therapy (with or without basal insulin) for a minimum of 3 months before the screening visit.
5. Subject is able and willing to self-monitor blood glucose level at home.
6. Subject has a body mass index (BMI) of ≥ 27 kg/m2 and ≤ 45 kg/m2.
7. Subject has metabolic syndrome, having at least 3 of the 5 risk factors.

Exclusion Criteria:

1. Subject is using prandial insulin or pre-mixed insulin in addition to oral hypoglycaemic agents for blood glucose control.
2. Subject is taking basal insulin dose > 1.0 U/kg/day.
3. Subject has recent or on-going infection requiring systemic treatment with an anti-infective agent within 30 days before screening.
4. Subject has a history of pancreatitis or diabetic ketoacidosis.
5. Subject has had at least one episode of severe hypoglycaemia in the past 12 months.
6. Subject has evidence of significant cardiovascular disease within 3 months before screening.
7. Subject has an estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2.
8. Subject has uncontrolled hypertension.
9. Subject has a diagnosis of rheumatic or inflammatory disease; or other autoimmune or inflammatory disease.
10. Subject is concurrently taking and plans to routinely continue taking anti-inflammatory medications during the study.
11. Subject is currently using medications for the indication of (or at the doses indicated for) weight loss.
12. Subject has significantly elevated liver enzyme levels.
13. History of malignancy of any organ system, treated or untreated, within the past 5 years other than basal or squamous cell skin cancer.
14. Subject has a history of chronic alcohol or other substance abuse.
15. Subject has a history of an allergic reaction to PBI-4050 or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of PBI-4050 400 mg, 800 mg, and 1200 mg as assessed by the number of subjects with abnormal laboratory values and/or adverse events that are related to treatment | 4 months
  Number of subjects with abnormal laboratory values and/or adverse events that are related to treatment
To evaluate the efficacy of PBI-4050 400 mg, 800 mg, and 1200 mg | 3 months
  Change from baseline on HbA1c levels

SECONDARY OUTCOMES:
Change from baseline on diabetic biomarkers | 3 months
  % reduction and/or increase of diabetic biomarkers such as fasting glucose, fasting insulin, fasting C-peptide
Change from baseline on pro-inflammatory/inflammatory biomarkers | 3 months
  % reduction and/or increase of biomarkers such as IL-6, IL-18, adiponectin
To evaluate the effect of PBI-4050 on frequency of hypoglycaemia events | 3 months
  Frequency of hypoglycaemia events

CONTACTS AND LOCATIONS:
Overall Officials: John Moran, MD, Study Chair — ProMetic Life Sciences Inc.
Locations (11):
- Canada (11):
  - C-Health, Edmonton, Alberta
  - Omnispec Clinical Research, Mirabel, Quebec
  - LMC Clinical Research Inc., Barrie
  - C-health - C-endo Division, Calgary
  - Centre de recherche clinique de Laval, Laval
  - Institut de Recherches Cliniques de Montreal (IRCM), Montreal
  - LMC Clinical Research Inc., Montreal
  - Manna Research, Québec
  - Synergy Medical Clinic, Sherwood Park
  - Manna Research, Toronto
  - Manna Research, Vancouver

IPD SHARING:
Plan to Share IPD: No